CLINICAL TRIAL: NCT00876369
Title: Vitamin D Levels in Subjects With Chronic Urticaria and Angioedema
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0045-09-EP
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Urticaria; Angioedema
Keywords: urticaria; angioedema; vitamin D; allergy
MeSH Terms: conditions — Urticaria; Angioedema; Hypersensitivity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Urticaria/Angioedema: Subjects with chronic urticaria and/or angioedema
- allergy control: Subjects with physician diagnosed allergic rhinitis

SUMMARY:
The objective of this study is to perform an exploratory analysis to determine if a possible relationship between vitamin D and chronic urticaria and/or angioedema exists. The study hypothesis is that vitamin D deficiency is associated with chronic urticaria and/or angioedema.

DETAILED DESCRIPTION:
The purpose of the research protocol is to perform a pilot study to determine the levels of 25-hydroxy vitamin D (25OHD), the storage form of vitamin D, in subjects with chronic urticaria and angioedema. Vitamin D is recognized as a key element in the regulation of the innate and adaptative immune system, and deficiencies of vitamin D could play an important role with inflammatory skin conditions such as chronic urticaria and angioedema.

Vitamin D deficiency has been implicated in contributing to the pathogenesis of skin inflammatory disorders including atopic dermatitis, rosacea and psoriasis. Deficiencies in vitamin D have recently been speculated to be associated with anaphylaxis diagnosis and treatment. The role of vitamin D in other allergic disorders such as allergic rhinitis is not clear. Chronic urticaria and angioedema (CUA) is a debilitating allergic disorder defined as recurrent urticaria and/or angioedema on a regular basis for greater than 6 weeks. The etiology of this disorder is largely unknown, but occurs predominately in females and can be associated with autoimmunity and thyroid disease. Vitamin D could potentially have an important role in the pathogenesis and treatment of CUA, but there are no studies to date examining the potential association of CUA and 25OHD levels.

This pilot study seeks to recruit two groups of adult subjects (ages 19 and up): 1) Control allergy group: subjects with physician-diagnosed allergic rhinitis, and 2) Subjects with physician-diagnosed chronic urticaria and/or angioedema. Subjects in the 2 groups will answer a questionnaire to collect information regarding demographics, vitamin D supplementation, previous diagnostic tests, current medications, and also a validated Dermatology Life Quality Index (attached). Other information will be obtained as available from the medical record: weight, height, body mass index (BMI), thyroid stimulating hormone (TSH), free thyroxine (T4), thyroid autoantibodies, urticaria autoimmune testing (autologous serum skin test, CD203c results), anti-nuclear antibody (ANA) and allergy skin prick testing. These stated tests are drawn for the evaluation of subjects with CUA. All subjects will have blood draw for 25OHD levels, and the levels will be compared between the 2 groups. It has been previously reported that approximately 15-30% of healthy populations are deficient in Vitamin D. There is no intervention component. Subjects will receive the 25OHD results, but no further follow-up is planned.

The objective of this pilot study is to perform an exploratory analysis to determine if a possible relationship between 25OHD and CUA exists, and to determine power calculations for a larger study. Finally, information regarding Vitamin D may be beneficial in determining potential contributing factors and also in the treatment of subjects with CUA.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1: subjects with physician-diagnosed allergic rhinitis. Allergic rhinitis is defined by clinical symptoms of sneezing, runny nose, nasal congestion and evidence of IgE-mediated disease (allergy skin prick test positive or radioallergosorbent test [RAST] positive to environmental inhalants such as trees, grasses, weeds, animal dander, molds, dust mite, cockroach).
2. Group 2: subjects with physician-diagnosed chronic urticaria and/or angioedema (CUA). CUA is defined by having urticarial wheals (hives) and/or angioedema (dermal swelling) on a daily or almost daily for more than 6 weeks.

Exclusion Criteria:

1. They are not capable of answering the questionnaire.
2. They are diagnosed with hereditary angioedema. Hereditary angioedema is a genetic disorder, autosomal dominant, of the C1 esterase inhibitor protein. These subjects will be excluded as the etiology of their disease is known.
3. Pregnant or lactating women. All child-bearing women will be asked (verbally and on the questionnaire) if they are pregnant or lactating. If they answer yes, they will be excluded. As there is no risk or harm to the pregnant or lactating woman, a urine pregnancy test will not be used.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects at subspeciality clinic (allergy/immunology) at tertiary care medical center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2009-12-11 (Actual); Study Completion 2009-12-11 (Actual)

PRIMARY OUTCOMES:
Vitamin D levels | one measurement
  A one-time blood draw from participants in chronic urticaria and/or angioedema group and control allergic rhinitis group will compare 25-hydroxy vitamin D (25OHD) levels between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jill A Poole, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States